CLINICAL TRIAL: NCT01895283
Title: The Effect of a Bike Ergometer Training Program in Patients With Bethlem Myopathy
Brief Title: The Effect of Aerobic Exercise, on Fitness and Functional Muscle Strength, in Patients With Muscular Dystrophy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Christoffer Rasmus Vissing, BsC, Rigshospitalet, Denmark
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: H-2-2013-066
Record Dates: First submitted 2013-07-03; First posted 2013-07-10 (Estimated); Last update posted 2016-04-06 (Estimated); Status verified 2016-04

CONDITIONS: Bethlem Myopathy
Keywords: Aerobic training; VO2max; Bethlem myopathy
MeSH Terms: conditions — Bethlem myopathy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Moderate-intensity training (Experimental): Regular supervised moderate-intensity training on a bike ergometer, three times per week, for 30 minutes a total of 10 weeks.
  Interventions: Behavioral: Moderate-intensity training

INTERVENTIONS:
Behavioral: Moderate-intensity training — Training at 70% of VO2max, for 1/2 hour, three times weekly, for 10 weeks, on a bike ergometer.

SUMMARY:
Muscular dystrophy is a group of disorders that are characterized by progressive muscle weakening and loss of muscle mass, caused by defects in muscle proteins. Muscular dystrophy is almost always inherited disorders, and so far, no curative treatments exist.

Previous studies have shown that endurance training significantly improves fitness and self-assessed muscle function in a variety of muscular dystrophies. In this study, we wish to investigate whether patients with Bethlem myopathy (a specific form of muscular dystrophy) also benefit from endurance training.

The study consists of two test days, a 10-week training period and five blood tests.

Patients will be required to train, three times per week, for 10 weeks, on a bike ergometer with a specific training intensity, under pulse rate monitoring.

The training period will be flanked by two test days, where we will determine, and compare the patients' muscle strength and fitness level, from before to after the training program. The patients conditioning level will be determined from a 15 minute cycle ergometer test and patients will undergo three functional tests to determine their functional muscle strength.

We will as a safety measure analyze blood tests before, during and after the training program for the muscle enzyme creatine kinase (an indicator of muscle damage) and through adverse effects as reported by patients during weekly telephone-consultations with the Principal investigator.

We anticipate, that Bethlem myopathy patients will have a similar rise in fitness level and functional muscle strength, as that seen in patients with other forms of muscular dystrophy, who undertake a similar training program.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Bethlem myopathy

Exclusion Criteria:

* Patients with disorders that would confound the interpretation of the effect from training (cardiomyopathy, pregnant women, etc.)
* Patients who are deemed mentally unfit for cooperation with the training program

Ages: 16 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2013-09; Primary Completion 2014-12 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Maximal oxygen uptake (VO2max) | after 10 week bike ergometer training program
  VO2max will be determined during an incremental bike test to exhaustion. VO2max is a physiological measure of physical fitness. VO2max relies on a persons ability to supply and consume oxygen ("energy") in muscle tissue.

SECONDARY OUTCOMES:
Functional muscle strength | After completion of a 10 week training program
  Functional muscle strength will be determined by performance in three functional tests: a five-repetition-sit-to-stand-test, a 6 minute walk test and a 14 step stair test.
Muscle strength determined by dynamometry | After completion of a 10 week training program
Self-assessed improvements in muscle function | After completion of a 10 week training program
Self-assessed improvements in incidence of problems that are related to inactivity (in patients who are confined to a wheel-chair) | After a 10 week training program

OTHER OUTCOMES:
Safety | During a 10 week training program
  The safety of undertaking a 10-week training program will be determined by analyzing reports of adverse effects faced during the training program, and by interpretation of Creatine Kinase levels measured before, during and after the training program.

CONTACTS AND LOCATIONS:
Overall Officials: Christoffer R Vissing, BsC, Principal Investigator — Rigshospitalet, Neuromuscular Research Unit
Locations (1):
- Rigshospitalet, Neuromuscular Research Unit, section 3342, Copenhagen, Denmark